CLINICAL TRIAL: NCT05644756
Title: IMPACT Center Signature Project 1, "Novel Methods for Implementing Measurement-Based Care for Youth in Low-resource Environments", is Embedded Within IMPACT Center P50 Entitled: Optimizing Evidence-Based Practice Implementation for Clinical Impact: the IMPACT Center.
Brief Title: Novel Methods for Implementing Measurement-Based Care for Youth in Low-resource Environments
Acronym: NIMBLE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Brown University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1943932-2; P50MH126219 (NIH)
Record Dates: First submitted 2022-11-18; First posted 2022-12-09 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Mental Health
Keywords: Youth Mental Health; Improving Measurement-based Care; Community Mental Health Centers; Implementation Science
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Measurement Based Care Implementation (Other): Four community mental health clinics located in Washington state will receive trainings on how to implement Measurement Based Care (MBC) in their clinics. We are creating implementation plans to improve therapists' use of measurement-based care.
  Interventions: Behavioral: IMPACT Methods to Identify and Prioritize Determinants (Challenge I), Challenge and Match strategies to Prioritized Determinants (Challenge II)

INTERVENTIONS:
Behavioral: IMPACT Methods to Identify and Prioritize Determinants (Challenge I), Challenge and Match strategies to Prioritized Determinants (Challenge II) — IMPACT Center developed two methods for identifying determinants that involved providers, staff, and youth at community mental health centers in site visit 1: Rapid Ethnographic Assessment, Design Probes. Then, practice partners engage in a facilitated group activity to rate the criticality, chronicity, and ubiquity of the list of determinants in Site Visit 2. Finally, practice partners engage in a third site visit where they create Causal Pathway Diagrams that allow them to match strategies to prioritize determinants and create Implementation Plans.

SUMMARY:
This study will visit 4 community mental health clinics in Washington state and work with clinic staff to find out if staff are regularly evaluating clinical outcomes using questionnaires (which is also called measurement-based care or MBC). The study team will partner with clinic staff to find out what makes using questionnaires difficult and then plan to improve the use of questionnaires. The study activities will include trainings, interviews, collaborative discussions, and interactive activities.

DETAILED DESCRIPTION:
Rapid Ethnographic Assessment (REA). REA will be conducted over 2-day site visits at each clinic, following a kickoff training on the principles of MBC. This team will conduct ethnographic observations on both days, using primarily unobtrusive techniques on Day 1, documenting observations of activities (e.g., clinician documentation), interactions (e.g., client check in), and events (e.g., staff meeting) using written and audio-recorded field notes. The investigators will interview staff for responses to the "example" question (for instance, "Could you show me how you use MBC in your work and describe what you are doing?") described above. The investigators expect up to 30 interviews per clinic: 30-45 minutes for therapists, 15 minutes for staff. The investigators will synthesize learnings from observations, interviews, and surveys in a debriefing session, using notes to generate a list of unique barriers. Day 2 will be focused observations of therapists shadowed by team members to document, track, and note the duration and location of activities, guided by barriers identified in the evidence review and Day 1 learnings. The investigators will conduct semi-structured, focused interviews based on Day 1 learnings, with therapists (therapists, supervisors, psychiatrists) and staff (up to 30). Day 2 interviews will be longer (15-30 minutes), audio recorded.

Design Kits. To complement REA and collect real-time data from therapists and youth, at the end of site visits, the investigators will leave design kit materials including disposable cameras, journals, pens and prompts to use to describe using MBC by taking pictures, make diary entries, draw maps, and record images. The investigators will ask therapists (5-8 per clinic) to participate.

Barrier Prioritization. The investigators will engage 5-8 therapists and/or staff in the prioritization activity for a 2-hour facilitated group activity. The activity will occur in-person (Site Visit 2) but could be delivered virtually if needed. Barriers identified through the rapid evidence review, rapid ethnographic assessment, and design kits (50+ expected) will be prioritized using a participant-engaged method.

Causal Pathway Diagramming. For each clinic, the investigators will develop Causal Pathway Diagrams (CPDs) for the top 3 prioritized barriers. The goal is to assess how well each implementation strategy is matched to a prioritized barrier, based on its mechanism of action, and to clarify the causal chain of events that must take place to achieve MBC fidelity.

Focus Groups to Improve IMPACT methods. The investigators will engage partners in a semi-structured focus group to capture their experience engaging in all IMPACT Center methods in the 3 site visits to inform further toolkit refinement. A facilitator not previously engaged in any of the activities will conduct a 60-minute focus group to solicit reactions to all aspects of IMPACT's methods, including the steps and personnel requirements of each method, and their output (e.g., prioritized barriers; utility of the information captured in the CPDs).

AIM 2: Compare MBC fidelity post IMPACT Center methods deployment versus historical controls.

The clinician self-report measure is a simple, quick, and homegrown self-report tool based upon the Collect, Share, Act conceptualization of MBC fidelity. The creation of this survey was guided by a need for something brief and pragmatic, and no self-report measures to our knowledge are (1) brief, (2) pragmatic, and (3) assess fidelity to the three main components of MBC. The survey asks clinicians to report (1) their approximate youth caseload in the last 6 months, and the percentage of youth patients with whom they have (2) collected data at least every two sessions, (3) shared data over the treatment course, and (4) acted on these processes to change the direction of treatment. Clinicians will complete this survey over REDCap. The study team will assess the internal reliability, concurrent validity, and convergent validity of the measure once data collection ends [41]. A copy of this measure is available from the first author.

The study will will present descriptive statistics to describe MBC fidelity at each of the three time points. The study will use a repeated measures analysis of variance to analyze whether fidelity to components of MBC changed from baseline (6 months after enrollment) to 3 months after active implementation, and finally 6 months after implementation.

ELIGIBILITY:
Inclusion Criteria:

* Aim 1: Co-create plans for optimizing Measurement Based Care (MBC) implementation for youth with comorbidities. Clinic staff/Therapists (N=180) across 6 CMHCs in Washington state.
* Aged 21+
* Working at a CMHC that is participating in the WA State CBT (Cognitive Behavioral Therapy) + Initiative.
* Aim 2: Compare MBC fidelity post IMPACT Center methods deployment (3-months and 6-months) versus pre-implementation. Clinic staff/Therapists (N=30) across 6 CMHCs in Washington.
* Must be aged 21+
* Working at a CMHC that is participating in the Washington State CBT (Cognitive Behavioral Therapy) + Initiative.

Exclusion Criteria:

* Aim 1: Clinic staff/Therapists: Unwilling to participate in study activities.
* Aim 2: Clinic staff/Therapists:
* Unwilling to respond to fidelity measure over REDCap

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-10-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-08-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben G Martinez, PhD, Study Director — Kaiser Permanente
Locations (1):
- KPWHRI, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martinez RG, Weiner BJ, Meza RD, Dorsey S, Palazzo LG, Matson A, Bain C, Mettert KD, Pullmann MD, Lewis CC. Study protocol: Novel Methods for Implementing Measurement-Based Care with youth in Low-Resource Environments (NIMBLE). Implement Sci Commun. 2023 Nov 28;4(1):152. doi: 10.1186/s43058-023-00526-z. PMID 38017522
- [Derived] Martinez RG, Cramer ER, Norris LA, Matson A, Lang C, Henrikson NB, Blasi PR, Palazzo LG, Hoopes AJ, Dorsey S, Weiner BJ. Short Report: Comparison of three methods for identifying implementation determinants to measurement-based care. Res Sq [Preprint]. 2025 Nov 19:rs.3.rs-7973723. doi: 10.21203/rs.3.rs-7973723/v1. PMID 41333394

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred at 3 distinct time points: October-November of 2022, June of 2022, and October of 2023. All recruitment was done in community mental health clinics.
Pre-assignment Details: For the first aim of the study (co-developing implementation plans), any member of participating community mental health center were invited to participate. After that, only therapists who served youth clients were included for the outcome data because they needed to be able to report on their use of outcome measures with youth clients. One clinic that enrolled clinic members later decided that they could not continue with the study, citing high waitlists and competing organizational priorities.
Groups:
- Measurement Based Care Implementation: Four community mental health clinics located in Washington state will receive trainings on how to implement Measurement Based Care (MBC) in their clinics. We created implementation plans to improve therapists' use of measurement-based care.
  IMPACT Methods to Identify and Prioritize Determinants (Challenge I), Challenge and Match strategies to Prioritized Determinants (Challenge II): IMPACT Center developed two methods for identifying determinants that involved providers, staff, and youth at community mental health centers in site visit 1: Rapid Ethnographic Assessment, Design Probes. Then, practice partners engage in a facilitated group activity to rate the criticality, chronicity, and ubiquity of the list of determinants in Site Visit 2. Finally, practice partners engage in a third site visit where they create Causal Pathway Diagrams that allow them to match strategies to prioritize determinants and create Implementation Plans.
  For aim 2, we evaluated whether the implementation plans had any effect on therapist's use of outcome questionnaires with their youth clients.
Period: Aim 1 Activities (Ethnography)
Arm/Group | Measurement Based Care Implementation
Started | 76
Completed (We originally planned to enroll patients in Aim 1 but were unsuccessful in recruiting patients, so no patients are included in this sample.) | 75
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Aim 2 Activities (Fidelity to MBC)
Arm/Group | Measurement Based Care Implementation
Started (This comment explains the discrepancy between the sample size of period 1 end and period 2 start. The period 1 rapid ethnography consisted of interviews with all manner of clinic staff: therapists, case managers, front desk staff, administrative staff. MBC fidelity evaluation (period 2) included only people who could report on using outcome questionnaires with clients, which includes only therapists and case managers.) | 35
Completed | 30
Not Completed | 5
Not completed — Lost to Follow-up | 5

BASELINE CHARACTERISTICS:
Population: This analysis population includes only youth-serving therapists, so it is a subset of the full sample.
Groups:
- Measurement Based Care Implementation: Four community mental health clinics located in Washington state will receive trainings on how to implement Measurement Based Care (MBC) in their clinics. We co-created implementation plans to improve therapists' use of measurement-based care by (1) identifying barriers and facilitators to MBC, (2) prioritizing barriers, and (3) co-developing an implementation strategy. The primary outcome of interest was whether the co-developed implementation strategies improved clinician's use of MBC (defined as % of youth clients administered measures) with youth clients.
  NOTE: Patients/clients were not enrolled in outcome measurement, as the study was primarily focused on whether implementation strategies improved clinicians use of measurement-based care (i.e., clinicians were the primary unit of analysis).
Arm/Group | Measurement Based Care Implementation
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Youth Clients Provided Outcome Questionnaires
Description: Aim 2 Therapists will report on the number of clinical outcome questionnaires administered to youth clients (the total number of outcome questionnaires per client used) before and after engaging in our researcher-driven implementation process.
Time Frame: We will assess at 6 (pre-implementation), 9 (3 months post-implementation), and 12 (6 months post-implementation) months after enrollment.
Measure: Mean (Standard Deviation); unit: number of youth clients given measures
Arm/Group | Measurement Based Care Implementation
Number analyzed (Participants) | 30
number of youth clients given measures
  Time 1 (pre-implementation) | 15.5 (14.7)
  Time 2 (3 months after implementation) | 16.7 (16.1)
  Time 3 (6 months after implementation) | 16.8 (15.8)
Statistical Analysis 1: Comparison: Measurement Based Care Implementation; Test type: Other — The primary analysis examined changes in measurement-based care (MBC) collection over time using ANOVA. The study was not designed as a superiority, non-inferiority, or equivalence trial; p > .01, ANOVA

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire implementation period of the study, so 12 months per clinic.
Arm/Group | Measurement Based Care Implementation
All-Cause Mortality (participants affected / at risk) | 0/76
Serious Adverse Events (participants affected / at risk) | 0/76
Other Adverse Events (participants affected / at risk) | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-04): https://cdn.clinicaltrials.gov/large-docs/56/NCT05644756/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT05644756/SAP_001.pdf